CLINICAL TRIAL: NCT00400374
Title: Phase I Study of Secondary Primary Tumor Prevention With Epidermal Growth Factor Receptor (EGFR), Tyrosine Kinase Inhibitor Erlotinib (OSI-774, Tarceva™), and Cyclooxygenase-2 (COX-2) Inhibitor (Celecoxib) in Early Stage (Stage I/II) Squamous Cell Carcinoma of Head and Neck
Brief Title: Secondary Primary Tumor Prevention With EGFR, OSI-774, and Cyclooxygenase-2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Genentech, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Dong Shin, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00021851; 5R01CA112643 (NIH)
Record Dates: First submitted 2006-11-15; First posted 2006-11-16 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Erlotinib Hydrochloride; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib, Celecoxib (Experimental)
  Interventions: Drug: Erlotinib; Drug: Celecoxib

INTERVENTIONS:
Drug: Erlotinib — Patients will be given Erlotinib (dose escalation from 50 mg, 75 mg, and 100 mg) once daily continuously for 6 months.
  Other Names: OSI-774; Tarceva
Drug: Celecoxib — Celecoxib, 400 mg, daily for 6 months.
  Other Names: SC-58635; Celebrex

SUMMARY:
This is a phase I study of second primary tumor prevention in early stage (stage I/II) patients diagnosed with squamous cell carcinoma of the head and neck (SCCHN).

DETAILED DESCRIPTION:
This is a phase I study of second primary tumor prevention in early stage (stage I/II) patients diagnosed with squamous cell carcinoma of the head and neck (SCCHN).

The study will evaluate the effect on cells and clinical response to study medications: Epidermal Growth Factor Receptor (EGFR), Tyrosine Kinase Inhibitor Erlotinib (OSI-774, Tarceva™), and Cyclooxygenase-2 (COX-2) Inhibitor (Celecoxib). The side effects of the medications will be assessed, and chemicals in the cells will be evaluated both before and after medication is administered that may show how the drugs work. This information will help researchers determine whether additional studies with these drugs should be conducted to determine if the drugs can help prevent pre-cancerous lesions from becoming cancerous.

SCCHN accounts for 5% of all cancer, and there is an incidence of approximately 37,200 new cases in the United States per year with 11,000 deaths. The five-year survival rate for patients with SCCHN in the United States and other developed countries is still poor, approximately 40%, comparable to the five-year survival rate in the 1970s despite advances in detection, surgery, radiation, and chemotherapy. Thus, a preventative approach before the development of invasive cancer or second primary tumors (SPTs) is highly desirable and novel strategies to reduce cancer incidence in SCCHN and other tobacco-carcinogen related malignancies are being pursued.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have, or have previously had, stage I (T1NO) or stage II (T2NO) squamous cell carcinoma of the head and neck.
* Tumor sites include oral cavity (buccal mucosal, gingival, floor of mouth, dorsal/ventral tongue, pharyngeal wall), oropharynx, larynx (glottis, supraglottis, subglottis, epiglottis) hypopharynx, paranasal sinus and nasal cavity.
* May have oral pre-malignant lesions (i.e., hyperplasia, dysplasia, carcinoma in situ) provided their Stage I or II disease has been definitively treated.
* Must have been free of disease for a minimum period of 8 weeks up to maximum of 3 years following completion of surgery and/or radiotherapy.
* Must have an Eastern Cooperative Oncology Group (ECOG)/Zubrod performance status of 0-1.
* Patients must be 18 years of age or greater.
* Female patients of childbearing potential must practice adequate contraception and have a negative pregnancy test (β-HCG).
* Must be able to swallow the Erlotinib and Celecoxib pills.
* Final eligibility for a clinical trial is determined by the health professionals conducting the trial.

Exclusion Criteria:

* Acute intercurrent illness or those who had surgery within the preceding 4 weeks unless they have fully recovered.
* History of previous malignancies other than squamous cell carcinoma of the head and neck unless the cancer was non-melanoma skin cancer.
* Participants who are pregnant or breast feeding.
* Documented history of coagulopathy and/or those taking warfarin or warfarin-derivative anticoagulants within 6 months of entry into the study.
* Hypertension not adequately controlled by medication as shown by a systolic ≥180 @ screening.
* Documented history of interstitial lung disease.
* Known connective tissue disease.
* Participated in a clinical trial of an investigational drug within 12 months prior to enrollment.
* Any active cardiovascular events including angina, unstable angina, palpitation, tachycardia, arrhythmia, or participant has had a recent cerebrovascular accident (stroke) or Myocardial Infarction (< 6 months).
* Any history of clinically significant ventricular arrythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de Pointes).
* Final eligibility for a clinical trial is determined by the health professionals conducting the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-08; Primary Completion 2012-12 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Define biologic dose of Erlotinib and Celecoxib in Erlotinib plus Celecoxib in patients with early stage (I/II) SCCHN. Improve overall survival rate by reducing SPTs and recurrence with combination of Erlotinib and Celecoxib. | 6 months

SECONDARY OUTCOMES:
Assess tolerability and toxicity associated with combination of Erlotinib and toxicity associated with combination of Erlotinib and Celecoxib for patients with early stage (I/II) SCCHN. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dong Shin, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Kim P, Saba NF, McCook-Veal A, Liu Y, Klein AM, Beitler JJ, Chen A, Khuri FR, Shin DM. Prospective Pilot Study of Second Primary Tumor Prevention With Erlotinib and Celecoxib in Early-Stage Squamous Cell Carcinoma of the Head and Neck: Long-Term Follow-Up. Head Neck. 2025 Sep;47(9):2594-2602. doi: 10.1002/hed.28178. Epub 2025 Apr 28. PMID 40296503